CLINICAL TRIAL: NCT04391881
Title: Oral Manifestation of COVID19
Brief Title: Oral Manifestation of COVID 19 Patient: A Cross Sectional Study on Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, Lecturer at conservative department, Cairo University
Other Study IDs: 54678
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Oral Health and COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The oral manifestation of COVID 19 that could help in the diagnosis of patient

DETAILED DESCRIPTION:
Oral ulceration,oral lesion,sensitivity that has been reported by patient tested positive for COVID 19

ELIGIBILITY:
Inclusion Criteria:

* Tested COVID positive
* No other chronic disease that has oral manifestation
* Above 18

Exclusion Criteria:

* Children
* Patient with no COVID positive

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Egyptian population tested COVID positive either hospitalized or not
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Oral manifestation | 1month
  The presence or absence or oral manifestation like ulcer burning sensation..will be measured by yes or no using a list of question

CONTACTS AND LOCATIONS:
Overall Officials: Dina Mounir Elkady, Principal Investigator — Lecturer at cairo ubiversity
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided